CLINICAL TRIAL: NCT01475903
Title: Assessment of Nutritional Consequences of Sleeve Gastrectomy
Acronym: ERNEST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0093; 2010-A00406-33
Record Dates: First submitted 2011-04-18; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
Keywords: Obesity; Sleeve gastrectomy; Nutritional impact; Vitamin deficiency
MeSH Terms: conditions — Obesity; Avitaminosis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- sleeve gastrectomy
  Interventions: Procedure: Longitudinal sleeve gastrectomy

INTERVENTIONS:
Procedure: Longitudinal sleeve gastrectomy — The main objective of this study is to assess during a 2-year prospective follow-up, the prevalence of nutrient deficiencies in patients undergoing a longitudinal sleeve gastrectomy for morbid obesity

SUMMARY:
Bariatric surgery is now recognized as a procedure of choice for the treatment of morbid obesity, resulting in long-term effectiveness on weight loss and comorbidities. The two types of procedures, most often performed in Europe, are adjustable gastric banding (AGB), a purely restrictive reversible procedure, and gastric bypass (GBP), an irreversible procedure, which associates restriction and mild malabsorption. Longitudinal sleeve gastrectomy (LSG) is another bariatric procedure which tends to develop quickly. More recent, this technique is recognized in France by the High Authority of Health since 2008, consisting of fundus and greater curvature resection, removing 75 % the gastric volume, leaving a narrow gastric tube or "sleeve".

Although malabsorption does not occur in most bariatric procedures, micronutrient deficiencies are possible. GBP is known to induce nutritional and vitamin deficiencies concerning iron, calcium, vitamins B12, B9, D and proteins. Restrictive procedures have minor effects on normal physiological digestive processes but could lead to vitamin deficiency secondary to decreased nutrient intake and a tendency towards avoidance of certain types of food due to intolerance. Studies of nutritional complications of bariatric surgery concern essentially AGB, GBP and vertical banded gastroplasty (VBG) which is no longer performed in France. The nutritional impact of LSG remains to be evaluated. To date, data concerning evaluation of nutritional status from patients who underwent LSG are almost non-existent. Considering this type of surgical procedure, the investigators expect to observe essentially a deficiency in vitamin B12 and iron. Indeed, defined as a purely restrictive intervention, LSG consists of gastric fundus resection which is the site of intrinsic factor production, itself necessary for vitamin B12 absorption. Moreover, decrease of hydrochloric acid production and potential vomiting caused by gastric resection can alter iron absorption.

In view of the increasing popularity of this surgical technique, assessment of the nutritional consequences of longitudinal sleeve gastrectomy seems to be necessary.

DETAILED DESCRIPTION:
Bariatric surgery is now recognized as a procedure of choice for the treatment of morbid obesity, resulting in long-term effectiveness on weight loss and comorbidities. The two types of procedures, most often performed in Europe, are adjustable gastric banding (AGB), a purely restrictive reversible procedure, and gastric bypass (GBP), an irreversible procedure, which associates restriction and mild malabsorption. Longitudinal sleeve gastrectomy (LSG) is another bariatric procedure which tends to develop quickly. More recent, this technique is recognized in France by the High Authority of Health since 2008, consisting of fundus and greater curvature resection, removing 75 % the gastric volume, leaving a narrow gastric tube or "sleeve".

Although malabsorption does not occur in most bariatric procedures, micronutrient deficiencies are possible. GBP is known to induce nutritional and vitamin deficiencies concerning iron, calcium, vitamins B12, B9, D and proteins. Restrictive procedures have minor effects on normal physiological digestive processes but could lead to vitamin deficiency secondary to decreased nutrient intake and a tendency towards avoidance of certain types of food due to intolerance. Studies of nutritional complications of bariatric surgery concern essentially AGB, GBP and vertical banded gastroplasty (VBG) which is no longer performed in France. The nutritional impact of LSG remains to be evaluated. To date, data concerning evaluation of nutritional status from patients who underwent LSG are almost non-existent. Considering this type of surgical procedure, the investigators expect to observe essentially a deficiency in vitamin B12 and iron. Indeed, defined as a purely restrictive intervention, LSG consists of gastric fundus resection which is the site of intrinsic factor production, itself necessary for vitamin B12 absorption. Moreover, decrease of hydrochloric acid production and potential vomiting caused by gastric resection can alter iron absorption.

In view of the increasing popularity of this surgical technique, assessment of the nutritional consequences of longitudinal sleeve gastrectomy seems to be necessary.

MAIN OBJECTIVE

The main objective of this study is to assess during a 2-year prospective follow-up, the prevalence of nutrient deficiencies in patients undergoing a longitudinal sleeve gastrectomy for morbid obesity

Obesity, defined by a body mass index (BMI) higher than 30 kg/m2, is a chronic metabolic disease the prevalence of which reaches epidemic proportions. Obesity increases the risk of hypertension, diabetes, and atherosclerosis, all risk factors for the leading cause of death worldwide-cardiovascular disease. Moreover, obesity can lead to obstructive sleep apnea, osteoarthritis, non-alcoholic fatty liver disease, cancer, etc…(Fried 2007). It represents one of society's major public health problems in (WHO 2000).

The treatment of obesity is primarily a medical matter. A multidisciplinary approach is recommended with nutritional, dietary and psychological follow-up. It requires a modification of life-style and long-term support. However, the long-term results of conventional medical therapy are disappointing, especially for morbid obesity. Bariatric surgery is now recognized as a procedure of choice for the treatment of morbid obesity. It's role in the therapeutic strategy is justified by long-term effectiveness on weight loss and comorbidities associated with high body mass index.

There are two types of bariatric procedures:

* Restrictive procedures, consisting of a reduction of the stomach volume : vertical banded gastroplasty (VBG), adjustable gastric banding (AGB), sleeve gastrectomy (SG)
* And combined procedures (restrictive and malabsorptive) : gastric by-pass and biliopancreatic diversion (BPD) with or without duodenal switch (DS).

The two types of procedures most often performed in Europe are AGB et GBP (Coupe 2009). VBG is tending to disappear in France, and biliopancreatic diversion (BPD), with or without duodenal switch (DS) is a complex procedure that is reserved for only very specific situations (Ziegler 2009).

Sleeve gastrectomy is a relatively new bariatric procedure. It was initially introduced as either the restrictive component of BPD-DS or the first step of a staged approach for weight loss. In the latter, super-obese patients with increased operative risks undergo SG to initiate enough weight loss to allow for a second stage gastric bypass or BPD-DS. It has been recently used as a definitive bariatric surgery procedure following reports of significant reduction in BMI and comorbidities. It is recognized in France by the High Authority of Health since 2008. SG is a laparoscopic bariatric procedure, in which the fundus and the greater curvature of the stomach are removed, leaving a narrow gastric tube or "sleeve" (Hakea 2009). Because of this partial gastrectomy, SG also affects ghrelin secretion which is an orexigenic hormone. These changes in the concentration of gut peptides induce a loss of appetite. The acceleration of the gastric emptying could also participate in weight loss (Ankar 2008). The advantages of sleeve gastrectomy reside in a lower rate of complications compared with BPG due in particular to the absence of implanted devices, the conservation of digestive continuity and the absence of malabsorption (Gums 2007). In terms of weight loss, the gastric by-pass appeared the most effective, followed by the sleeve gastrectomy, then the adjustable gastric ring. According to a recent meta-analysis, the loss of weight expressed in percentage of reduced excess weight was 61,6 % for the BPG and 47,5 % for the GB within 2 years of the procedure (Buchwald 2004). Concerning the sleeve gastrectomy, a review of the literature comprising 15 studies and including 646 patients, shows evidence of a reduction of excess weight of 49 % and 56 % after 6 months and 1 year respectively with a resolution of co-morbidity such as arterial high blood pressure and type 2 diabetes, from 60 to 100 % (Gums : 2007). The data on long-term follow-up is less well documented.

The risk of nutritional deficiencies depends on the percentage of weight loss and the type of surgical procedure performed The nutritional deficits observed after gastric surgery can be explained by various mechanisms according to the technique used. T BPG, which is both restrictive and malabsorptive surgery, is frequently at the origin of nutritional and vitamin deficiencies essentially concerning proteins, iron, calcium, vitamins B12, B9 and D. In contrast, in the absence of malabsorption, the nutritional deficits induced by AGB are less pronounced and particularly linked to contribution deficiencies due to vomiting, food aversions and modification of food supply .Studies evaluating the nutritional status of patients before and after surgery are scarce and prevalency of the reported deficits varies greatly according to the population studied, the type of surgery used, the systematic prescription or not of vitamin complements, and the duration of follow-up.

The most frequent deficit is the deficiency in vitamin B12, found in 1/3 of the one year follow up BPG patients (Malone 2008). Folate deficiency (vitamin B9) is also frequent, arising in 20 % of cases (Pournaras 2009). Both are at the origin of macrocytic anaemia, leucopenia, thrombopenia and glossitis. Sometimes irreversible neurological affections can also arise in the case of B12 deficiency. The effects of bariatric surgery on vitamin D and calcium are rarely specified in the long term, but it is important to note that it is not rare to observe vitamin D deficiencies pre-existent to surgery affecting between 21 and 57 % of obese subjects according to certain studies, (Toh 2009, Hamoui 2004), responsible for an increase in osseous fragility and secondary hyper-parathyroidism. The patients most at risk of osteomalacia would be the ones whose BMI is over 50, menopause women, patients having undergone a massive loss of weight after surgery and patients deficient in vitamin D prior to surgery (Malone 2008). Bariatric sideropenic anaemia is also frequent after surgery whether restrictive or malabsorptive, affecting 5 to 10 % of the subjects in most of the studies and as many as 74 % according to one study (Sadoul 2007). It is linked to contribution deficiency due to decreased consumption of meat, in the case of malabsorption (BPG) but also due to lack of production of gastric hydrochloric acid which allows the conversion of the ferrous iron foodstuffs to ferric iron, which is the absorbable form. Other vitamin deficiencies were reported, in particular the deficit in vitamin B1 (or thiamine) , essentially due to vomiting because of the gastric limitation, and which can be revealed by an intravenous drip of thiamine-free glucose. Vitamin B1 deficiency, although rather rare, is potentially serious because of neurological damage such as the sometimes irreversible Gayet-Wernicke's syndrome, (Poitou 2008; Morel 2008). Deficits in liposoluble vitamins A, E and K are exceptional except in the case of serious malabsorption induced by bilic-pancreatic diversion and duodenal switch. Zinc, magnesium and selenium deficiencies are also described but remain rare and originate mostly through exoskeleton or cutaneous disorders but cases of cardiomyopathy by selenium deficiency was also reported .

To date, recommendations on the optimal vitamin supplementation to be prescribed according to the method of surgery used are not clearly defined. According to recent recommendations of the HAS for the surgical care of adult obesity, " the medical and surgical follow-up must emphasize the prevention of, and the detection of, vitamin or nutritional deficiency including the identification of clinical (in particular neurological) and biological symptoms of undernutrition or vitamin deficiency. A systematic multivitamin supplementation must be established after malabsorptive surgery (multivitamins, vitamin D, calcium, iron and vitamin B12). " However, certain authors report deficiencies in spite of systematic prescription of multivitamin supplements after by-pass surgery .Data on the prescribed doses, controls, or even the preliminary nutritional state before surgery remains badly specified. On one hand, the rarity of prospective studies evaluating these parameters explains the difficulty in estimating these nutritional complications. On the other hand, the various studies listed refer essentially to gastric by-pass, the adjustable gastric ring, and the calibrated vertical gastroplasty which is tending to disappear. The impact of the sleeve gastrectomy on the nutritional state of the patients remains to be specified. To date, data concerning the vitamin and nutritional evaluation of patients operated by sleeve gastrectomy is almost non-existent. A recent review of the literature did not reveal any nutritional recommendations specifically for sleeve gastrectomy mostly due to the very small number of studies available. An American team studied the evolution of the nutritional assessment in the case of sleeve gastrectomy but the parameters studied were limited to albumin, haemoglobin and calcium. A decrease of the haemoglobinaemia was objectivized to 5 of 36 patients followed during 1 year .An Australian team also retrospectively estimated prevalency of nutritional deficiencies after bariatric surgery, but the data concerning sleeve gastrectomy is not significant considering the large number of patients lost sight of in 1 year (> 80 %) (Toh 2009).

The growing interest in LSG as a surgical procedure for managing morbid obesity requires further investigation of it's metabolic consequences.

In view of the increasing popularity of this surgical technique the evaluation of the nutritional repercussions of sleeve gastrectomy appears indispensable. If the investigators consider the surgical aspect of this procedure, the investigators would expect to observe a deficiency in vitamin B12 and iron. Indeed, defined as a purely restrictive procedure, the sleeve gastrectomy consists of the resection of the gastric fundus, the seat of production of the intrinsic factor, itself necessary for the absorption of vitamin B12. Moreover, the decrease in production of hydrochloric acid and the potential vomiting caused by the vast gastric resection can potentially have an effect on the absorption of iron. The study proposed here aims to make a prospective follow-up of the nutritional and vitamin assessment of obese patients operated by sleeve gastrectomy at the University Hospital of Clermont-Ferrand. Every patient will receive a clinical and biological assessment including the dosages of vitamins and trace elements prior to surgery then after 3, 6, 12, 18 and 24 months. The effect of sleeve gastrectomy on the nutritional status of the operated patients will thus be evaluated with a view to answering the question: Is sleeve gastrectomy a purely restrictive surgical technique ?

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Initial BMI = 35
* Proposition of a sleeve gastrectomy during a multidisciplinary consultation
* Bariatric surgery procedure carried out at the University Hospital of Clermont- Ferrand.
* Patient covered by the national health insurance scheme
* Patient having read, understood and signed the information sheet and the consent form

Exclusion Criteria:

* History of pathology or major surgical procedure which could interfere with the nutritional state and other study parameters (cancer, DID, digestive pathology, infectious or inflammatory disease)
* Pregnant or breast-feeding women
* Existence of cognitive disorders which could interfere with compliance of the study
* Person deprived of judicial or administrative freedom
* Participation in another study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: defined population
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
micro nutritional status of patients undergoing sleeve gastrectomy | at 3, 6, 12, 18 and 24 months after intervention

SECONDARY OUTCOMES:
physical composition measured by impedancemetry | at 3, 6, 12, 18 and 24 months
arterial blood pressure | at 3, 6, 12, 18 and 24 months
HOMA test | at 3, 6, 12, 18 and 24 months
lipid assessment | at 3, 6, 12, 18 and 24 months
arthropathy estimated clinically | at 3, 6, 12, 18 and 24 months
questionnaire SF-36 | at 6 months after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Julie LEGER-GUIST'HAU, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France